CLINICAL TRIAL: NCT00945087
Title: Experimental Phage Therapy of Drug-resistant Bacterial Infections, Including MRSA Infections
Brief Title: Experimental Phage Therapy of Bacterial Infections
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Immunology and Experimental Therapy of the Polish Academy of Sciences (Other)
Other Study IDs: OTF-1
Record Dates: First submitted 2009-07-21; First posted 2009-07-23 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-08

CONDITIONS: Bacterial Infections
Keywords: bacteriophage; bacteriophage preparation; bacterial infection; antibiotic-resistant infection; multidrug-resistant bacteria; MRSA
MeSH Terms: conditions — Bacterial Infections

INTERVENTIONS:
Other: Bacteriophage preparation — Bacteriophage lysates or purified phage formulations containing phages lytic for Staphylococcus, Enterococcus, Pseudomonas, Escherichia, Klebsiella, Proteus, Citrobacter, Acinetobacter, Serratia, Morganella, Shigella, Salmonella, Enterobacter, Stenotrophomonas, or Burkholderia strains isolated from a patient used for oral, rectal and/or topical application.
  Other Names: Phage preparation, bacteriophage formulation

SUMMARY:
The primary purpose of this experimental therapy is to treat, with the aid of bacteriophages, patients with non-healing postoperative wounds or bone, upper respiratory tract, genital or urinary tract infections in whom extensive antibiotic therapy failed or the use of the targeted drug is contraindicated.

DETAILED DESCRIPTION:
Bacterial infections of different tissues and organs that prove incurable by antibiotics are a serious clinical problem. Bacteriophages (phages) are bacterial viruses which attack, multiply within, and then destroy bacteria. They can efficiently destroy bacteria which have acquired resistance to antibiotics and which cause life-threatening infections. The method of treating bacterial infections using phages has been known since the beginning of the 20th century. This experimental treatment enables the use of phage preparations under the rules of a therapeutic experiment (on the basis of the respective Polish regulations) in cases where no effective available therapy exists or the use of the targeted drug is contraindicated. It is not a research study.

The bacteriophage preparations which are used in the treatment procedures contain phages from the Bacteriophage Collection of the Institute of Immunology and Experimental Therapy of the Polish Academy of Sciences in Wrocław. For each patient only specific formulations of single phage or a phage mixture that are active against the pathogenic bacterial strain or strains isolated from the patient are used for the treatment.The isolation of live bacterial pathogen from the patient is necessary to carry out a phage-typing procedure to determine if the preparation of an active formulation is possible which is a prerequisite for receiving the treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or over.
* Men and women of reproductive age must use contraception during and one month after the therapy. Women of reproductive age must have negative result of a pregnancy test before beginning of the treatment.
* Signed informed consent.
* Antibiotic therapy-resistant, chronic, symptomatic bacterial infection of the skin, subcutaneous tissue, bone, bone marrow, joints, fistulas, wounds, bedsores, genital and/or urinary tract, digestive tract, middle ear, sinuses, tonsils, upper and lower respiratory tract, or a state in which a targeted antibiotic therapy is impossible to carry out due to other medical reasons.
* A putative pathogenic bacteria such as Staphylococcus, Enterococcus, Escherichia, Citrobacter, Enterobacter, Klebsiella, Shigella, Salmonella, Serratia, Proteus, Pseudomonas, Stenotrophomonas, Acinetobacter, Burkholderia, or Morganella present in the site of the said infection as confirmed by the result of microbiological culture.
* Ineffective antibiotic therapy of said infection and/or antibiogram-confirmed multidrug resistance of a putative pathogenic bacteria such as Staphylococcus, Enterococcus, Escherichia, Citrobacter, Enterobacter, Klebsiella, Shigella, Salmonella, Serratia, Proteus, Pseudomonas, Stenotrophomonas, Acinetobacter, Burkholderia, or Morganella.
* The presence in the Bacteriophage Collection of the Institute of Immunology and Experimental Therapy of the Polish Academy of Sciences of a phage able to lyse a bacterial strain cultured from a patient in the Bacteriophage Collection of the Institute of Immunology and Experimental Therapy of the Polish Academy of Sciences (positive result of a phage-typing procedure).

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Malabsorption syndrome, allergy to food or animal protein, or advanced hepatic insufficiency when it is impossible to apply the phage preparation using other route than oral.
* Allergy to components of phage preparations.
* A health condition which does not allow conducting the experimental therapy in the opinion of the qualifying physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej Górski, M.D. Ph.D., Study Director — Institute of Immunology and Experimental Therapy of the Polish Academy of Sciences
Locations (1):
- Phage Therapy Unit at the Institute of Immunology and Experimental Therapy of the Polish Academy of Sciences, Wroclaw, Poland

REFERENCES:
- [Result] Miedzybrodzki R, Borysowski J, Weber-Dabrowska B, Fortuna W, Letkiewicz S, Szufnarowski K, Pawelczyk Z, Rogoz P, Klak M, Wojtasik E, Gorski A. Clinical aspects of phage therapy. Adv Virus Res. 2012;83:73-121. doi: 10.1016/B978-0-12-394438-2.00003-7. PMID 22748809
- See also: Click here for more information about this study: Experimental phage therapy of drug-resistant bacterial infections, including MRSA infections (in Polish) — http://surfer.iitd.pan.wroc.pl/pl/OTF/
- See also: Bacteriophage research and therapy — http://surfer.iitd.pan.wroc.pl/en/Phages/